CLINICAL TRIAL: NCT00651495
Title: Activating Seniors to Improve Chronic Disease Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Foundation for Informed Medical Decision Making (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: G07-09-025; FIMDM 0096-1
Record Dates: First submitted 2008-03-28; First posted 2008-04-02 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: Healthy
Keywords: Decision aids; Seniors; Chronic disease management; Advance directives

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Participants receive a $50 financial incentive if they view at least 3 of 5 patient decision aids in a group screening.
  Interventions: Behavioral: Patient decision aids for chronic conditions
- 2 (Active Comparator): No financial incentive for watching patient decision aids in group screenings
  Interventions: Behavioral: Patient decision aids for chronic conditions

INTERVENTIONS:
Behavioral: Patient decision aids for chronic conditions — Videos providing comprehensive information about chronic disease management

SUMMARY:
Chronic diseases are the primary cause of morbidity and mortality for older Americans. Active patient participation in treatment decision-making has the potential to significantly improve outcomes in chronic disease care, but interventions to increase participation remain underused. Some studies have found that older individuals are less interested in participating in clinical decision-making, but other studies find that exposing patients to decision aids (PtDAs) increases their desire to take an active role in making decisions with their physicians. The present study targets hard-to-reach seniors by showing decision aids focused on chronic disease management in senior centers. Decision aids will be made available in two senior centers through a lending library and by conducting group screenings of the decision aids followed by moderated discussion of the content with participants. A randomized encouragement design will be used to test the effectiveness of a modest financial incentive on increasing seniors' participation in group screenings. The investigators will evaluate the effects of the intervention on seniors' decision-making role preferences, attitudes, perceived social norms and self efficacy for asking questions of their physician, health-related quality of life, physical activity, and changes in prescribed treatment regimens and self-care.

ELIGIBILITY:
Inclusion Criteria:

* At least 55 years old.
* Able to ambulate
* Able to complete self-administered surveys
* Able to speak and read English

Exclusion Criteria:

* Not willing to provide consent

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2008-04; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Decision-making role preferences | 20 weeks
Attitudes, perceived social norms and self efficacy for asking questions of a physician | 20 weeks

SECONDARY OUTCOMES:
Health-related quality of life | 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dominick L Frosch, Ph.D., Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - Culver City Senior Center, Culver City, California
  - Willowbrook Senior Center, Los Angeles, California

REFERENCES:
- [Result] Frosch DL, Rincon D, Ochoa S, Mangione CM. Activating seniors to improve chronic disease care: results from a pilot intervention study. J Am Geriatr Soc. 2010 Aug;58(8):1496-503. doi: 10.1111/j.1532-5415.2010.02980.x. Epub 2010 Jul 19. PMID 20662953